CLINICAL TRIAL: NCT07131865
Title: Effectiveness Analysis of Inpatient Geriatric Rehabilitation According to the Valensian Model
Brief Title: Comparison of the Functional Status, Psychosocial Aspects and Discharge Locations of Geriatric Patients Before and After Inpatient Geriatric Rehabilitation
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-00382; EKOS 25/028 (Other: Ethikkommission Ostschweiz (EKOS))
Record Dates: First submitted 2025-08-12; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Weak; Senile; Old Age; Debility; Movement Disorders; Quality of Life; Sarcopenia
Keywords: Rehabilitation; Geriatrics; Effectiveness; Frailty
MeSH Terms: conditions — Asthenia; Frailty; Movement Disorders; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to demographic change in Switzerland, the proportion of older people in the population is expected to increase. It is therefore important that people in old age remain in the best of health and maintain their independence for a long time.

To this end, the investigators would like to demonstrate the effectiveness of inpatient geriatric rehabilitation at the Valens clinics. This will be done by comparing independence, quality of life, physical and mental health, mobility and hand strength on admission and discharge.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were treated as inpatients at the Kliniken Valens Geriatric Rehabilitation according to ICF criteria between 2020 and 2023 will be included.
* Signed the general consent for the further use of their health-related data for research, version 1.2, dated November 18, 2019.

Exclusion Criteria:

* No written consent was provided.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Age greater than 65 years
  Presence of multimorbidity
Sampling Method: Non-Probability Sample
Enrollment: 753 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Classification of diagnosis into internal medicine, neurological, or orthopedic/surgical categories | At baseline (upon hospital admission and study enrollment)
  Number of participants with diagnoses are divided into 3 groups: internal medicine, neurology and orthopedic/surgical. The diagnoses are determined and documented at hospital admission based on prior clinical assessments, laboratory results, and imaging studies. They are classified into one of three categories:
  Internal medicine (e.g., cardiovascular, respiratory diseases), Neurological (e.g., stroke, neuropathies) or Orthopedic/surgical (e.g., fractures, joint disorders). This classification reflects the patient's primary diagnosis at the time of study enrollment.
Cumulative Health Rating Scale (CIRS) | At baseline (upon hospital admission and study enrollment)
  The Cumulative Illness Rating Scale is a tool used to measure the overall burden of chronic illnesses across multiple organ systems. Each system is rated from 0 (no problem) to 4 (severe problem), and the scores are added up to reflect a patient's total morbidity. It is commonly used in geriatrics to assess multimorbidity and help predict health outcomes.
Functional Independence Measure (FIM) | At baseline (upon hospital admission and study enrollment) and at discharge from the clinic after a stay of approx. 21 days
  The FIM assesses how independently a person can perform daily activities. It uses an 18-item scale covering motor and cognitive tasks, each rated from 1 (total assistance needed) to 7 (complete independence). The total score reflects the level of disability and the amount of assistance required for daily living. Higher scores mean greater independence.
Health-related quality of life (EQ5D-5VAS) | At baseline (upon hospital admission and study enrollment) and at discharge from the clinic after a stay of approx. 21 days
  The EQ-5D-5VAS is a brief, standardized questionnaire for measuring health-related quality of life. It consists of two parts Descriptive system: Assesses five dimensions-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression-each with five levels of severity, allowing patients to describe their health state precisely and Visual Analogue Scale (VAS): Patients rate their overall health on a scale from 0 (worst imaginable health) to 100 (best imaginable health), providing a quantitative self-assessment
Patient Reported Outcomes Measurement Information System - (PROMIS-10) | At baseline (upon hospital admission and study enrollment) and at discharge from the clinic after a stay of approx. 21 days
  It is a short, 10-item questionnaire that measures subjective physical and mental health from the patient's perspective. It covers areas like physical function, pain, fatigue, emotional distress and social health. It helps researchers understand how the patients are feeling in terms of both body and mind.
  Higher scores indicate better health.
Timed Up and Go Test (TUG) | At baseline (upon hospital admission and study enrollment) and at discharge from the clinic after a stay of approx. 21 days
  The Timed Up and Go (TUG) test is a simple test for assessing mobility and balance. The person stands up from a chair, walks three meters, turns around, walks back, and sits down again. The time required to complete the task is measured.
Grip strength measured by the Jamar Hand Dynamometer | At baseline (upon hospital admission and study enrollment) and at discharge from the clinic after a stay of approx. 21 days
  The Jamar Hand Dynamometer is a standardized instrument used to measure grip strength, which reflects the maximum force exerted by the hand muscles during a squeeze.
  The grip strength is an important functional outcome and indicator of overall muscle strength and physical health. It is a reliable, non-invasive, and easy-to-administer test that provides valuable information about the participant's muscular strength and functional status.
  Participants will be asked to squeeze the dynamometer handle with maximum effort for a few seconds. The device will record the force applied, reported in kilograms.

SECONDARY OUTCOMES:
Age of participants | At baseline (upon hospital admission and study enrollment)
  Participant age will be recorded in years at the time of study enrollment. Age is an important demographic variable used to characterize the study population and to analyze outcomes by age groups if applicable.
Gender of participants | At baseline (upon hospital admission and study enrollment)
  Participant gender will be recorded as male, female, or other at the time of study enrollment. Gender is a key demographic variable to describe the study population and analyze potential differences in outcomes.
Marital status of participants | At baseline (upon hospital admission and study enrollment)
  Marital status will be recorded at the time of study enrollment and categorized as single, married, divorced, widowed, or other. This demographic information helps to characterize the study population and may be used to analyze its influence on health outcomes.
Place of residence of participants | At baseline (upon hospital admission and study enrollment)
  Participants' place of residence will be recorded at the time of study enrollment. This information may include urban or rural status, region, or postal code. It helps to describe the study population and assess potential geographic influences on health outcomes.
Length of hospital stay | From the beginning of the study (at hospitalization and admission to the study) until discharge from the clinic after a stay of approx. 21 days
  The length of hospital stay will be recorded in days, calculated from the date of admission to the date of discharge. This measure reflects the duration of inpatient treatment and may be used to evaluate resource utilization and recovery time.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Stefan Bachmann, Prof. Dr. med., Study Chair — University of Bern, Kliniken Valens
Locations (1):
- Kliniken Valens, Rehazentrum Walenstadtberg, Walenstadtberg, St.Gallen, Switzerland